CLINICAL TRIAL: NCT05450146
Title: Trial-based Effectiveness and Cost-effectiveness of the Partner in Balance Intervention to Selfmanage Mild Dementia Via Blended eHealth Psycho-education and Behavioural Modelling for the Care Partner Coached by a Case Manager
Brief Title: Trial-based Effectiveness and Cost-effectiveness of the Partner in Balance Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: VU University of Amsterdam (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: METC 2021-2955; 80-85200-98-21039 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Dementia, Mild
Keywords: early-stage dementia; informal caregiver; informal care
MeSH Terms: conditions — Dementia; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partner in Balance (intervention group) (Experimental): Informal caregivers assigned to the intervention group will receive the 8-week online selfmanagement program "Partner in Balance" (Boots, 2018).
  Interventions: Other: Partner in Balance
- Usual/standard care (control group) (No Intervention): Participants in the comparison condition will continue to receive the care as usual.
  The control group will be shared with another collaborating study from the 'Vrije Universiteit of Amsterdam'), which has the same goals, applies the same inclusion criteria, applies the same study procedures, and obtains the same outcomes. This implies that the data of the participants recruited for the control group for this study will be shared with the collaborating study.

INTERVENTIONS:
Other: Partner in Balance — The "Partner in Balance" intervention (Boots, 2018) consists of 1) a face-to-face intake session with a care professional (casemanagers, dementia nurses or district nurses) to familiarize participants with the program, set goals, and select preferred module themes; 2) tailored online thematic modules, including psychoeducation, behavioral modeling, reflective assignments, set goals, and online messaging feedback with the care professional over 8 weeks; and 3) a face-to-face evaluation session with the care professional evaluating previously set goals.
  Arms: Partner in Balance (intervention group)

SUMMARY:
Rationale:

Informal care is one of the most important sources of care for dependent elderly people. The Partner in Balance (PIB) intervention aims to prepare and support informal caregivers for their caregiving tasks. Long-term cost-effectiveness evidence is required to support reimbursement decision-making on this PIB program. The investigators hypothesize that 1) caregiver self-efficacy in intervention arm PiB is higher compared to the control arm of usual care; 2) care costs of participants in intervention arm are lower compared to the control arm of usual care.

Objectives:

The investigators aim to answer the following research questions:

* What is the effect of PiB on caregiver self-efficacy compared to usual care?
* What is the effect of PiB on caregiver and person with dementia total care costs compared to usual care?
* What is the incremental cost-utility ratio of PiB compared to usual care?
* What is the annual budget impact of PiB compared to usual care?

Study design:

Pragmatic, cluster randomised controlled trial.

Study population:

Informal caregivers of people with early-stage dementia who are community-dwelling and are receiving little or no dementia-related formal ADL-care

Intervention: blended E-health informal caregiver support program with online psycho-education and behavioural modelling. It contains personalized goal setting, online modules with option for online communication with care professional, evaluation with care professional.

Main study parameters/endpoints:

Primary: self-efficacy. Cost-utility: EQ5D, RUD. Secondary: quality-of-life, caregiver burden

Data collection:

Measurements consist of questionnaires (total duration is approximately 1 hour; administered at home, via telephone, via email or other location if preferred by the participant; take place at baseline, 3, 6, 12 and 24 months).

ELIGIBILITY:
Inclusion Criteria:

* Subject is an informal caregiver of a person with early stage dementia.
* The caregiver provides support for a person with dementia who is diagnosed of dementia (self-reported or known by the recruiting organization) or underdiagnosed dementia (no formal diagnosis but symptoms of dementia)
* The caregiver provides support for a person with dementia who is not yet receiving formal care related to personal activities of daily living on account of his/her dementia more than two times a week (defined by receiving assistance from a paid worker by e.g., health or social care such as help with dressing/undressing, washing/bathing/showering, toileting, feeding/drinking, taking medication or attending day activity or day care centre).

Exclusion Criteria:

* The informal caregiver is participating in another trial with similar objectives as this research.
* The informal caregiver has a major mental or physical illness
* The informal caregivers' person with dementia has a major mental or physical illness.
* The dementia of the informal caregivers' person with dementia is caused by human immunodeficiency virus (HIV), acquired brain impairment, Down syndrome, chorea associated with Huntington's disease, or alcohol abuse.
* Informal caregiver is younger than 18 years old.
* Informal caregiver or person with dementia does not have a minimum understanding of Dutch language.
* Informal caregiver has no basic internet skills.
* Informal caregiver has no access to internet at home.
* Informal caregiver has not received the online cursus 'Partner in Balance' yet.
* Informal caregiver is not receiving a similar support program.
* The informal caregiver is not able to follow COVID19 instructions. Type of dementia (e.g., Alzheimer, vascular) will not be a selection criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy | 24 months
  The self-efficacy of informal caregivers measured by the Caregiver Self-efficacy Scale (CSES) (Fortinsky, 2002). The maximum and minimum answer scores range from 1 to 10 with higher scores indicating better outcomes.
Health-related quality-of-life | 24 months
  Health-related quality-of-life of the informal caregivers and persons with dementia measured by the EQ-5D-5L. The questionnaire is scored on a 5-point Likert scale.
Healthcare resource use | 24 months
  Healthcare resource use of the informal caregivers and persons with dementia measured by the Resource Utilization in Dementia (RUD) (Wimo, 2013).

SECONDARY OUTCOMES:
Depression and anxiety | 12 months
  Depression and anxiety of informal caregivers measured by the Hospital and Anxiety Depression Scale (HADS) (Bjelland, 2002). The questionnaire is scored on a 4-point Likert scale.
Quality of life (informal caregiver) | 24 months
  Quality of life of informal caregivers measured by the Investigating Choice Experiments for the Preferences of Older People CAPability measure for Older people (ICECAP-O) (Makai, 2015). The questionnaire is scored on a 4-point Likert scale.
Quality of life (person with dementia) | 24 months
  Quality of life of persons with dementia measured by the Quality of Life- Alzheimer's Disease scale (QOL-AD) (Logsdon et al., 2002). The questionnaire is scored on a 4-point Likert scale.
Experienced burden of informal care | 12 months
  Experienced burden of informal caregivers measured by the EDIZ ("Ervaren Druk door Informele Zorg" / experienced burden of informal care) (Pot, 1995). The questionnaire is scored on a 5-point Likert scale.
Participant characteristics | baseline
  Characteristics of the informal caregivers and persons with dementia collected by the TOPICS-MDS questionnaire to capture TOPICS-MDS:
  * demographic characteristics
  * relation between informal caregiver and person with dementia
  * perseverance time (informal caregiver)
  * instrumental and personal activities of daily living (person with dementia)
Cognitive status of the person with dementia as estimated by the informal caregiver | baseline
  Cognitive status of the person with dementia as estimated by the informal caregiver measured by a selection of the Quick Dementia Rating System (QDRS). The questionnaire is scored on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein de Vugt, professor, Study Director — Maastricht University
Locations (1):
- Alzheimer Centrum Limburg, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Boots LM, de Vugt ME, Withagen HE, Kempen GI, Verhey FR. Development and Initial Evaluation of the Web-Based Self-Management Program "Partner in Balance" for Family Caregivers of People With Early Stage Dementia: An Exploratory Mixed-Methods Study. JMIR Res Protoc. 2016 Mar 1;5(1):e33. doi: 10.2196/resprot.5142. PMID 26932438
- [Background] Boots LM, de Vugt ME, Kempen GI, Verhey FR. Effectiveness of the blended care self-management program "Partner in Balance" for early-stage dementia caregivers: study protocol for a randomized controlled trial. Trials. 2016 May 4;17(1):231. doi: 10.1186/s13063-016-1351-z. PMID 27142676
- [Derived] Osstyn SL, Handels R, Boots LMM, Balvert SCE, Evers SMAA, de Vugt ME. The effectiveness and health-economic evaluation of "Partner in Balance," a blended self-management program for early-stage dementia caregivers: study protocol for a cluster-randomized controlled trial. Trials. 2023 Jun 22;24(1):427. doi: 10.1186/s13063-023-07423-9. PMID 37349828